CLINICAL TRIAL: NCT03646877
Title: Mechanisms of Ozone-Induced Alterations in Efferocytosis and Phagocytosis
Acronym: MOZEPH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Tighe, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Robert Tighe, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PRO00100375; ES028829 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ozone (O3) (Experimental): The O3 level during the exposures will be 200 ppb, which has previously been used in human exposure studies without short or long term, untoward side effects (and comparable to peak levels attained during the summer in the Raleigh-Durham area of North Carolina) (REF - Bromberg review).
  Interventions: Drug: Ozone
- Filtered Air (FA) (Placebo Comparator): Control will be treadmill walk with filtered room air in chamber.
  Interventions: Other: Filtered Air

INTERVENTIONS:
Drug: Ozone — Subjects will perform alternating 15 minutes rest with 15 minutes treadmill walk exercise periods for 135 minutes in while breathing Ozone (O3).
  Other Names: O3
  Arms: Ozone (O3)
Other: Filtered Air — Subjects will perform alternating 15 minutes rest with 15 minutes treadmill walk exercise periods for 135 minutes in while breathing filtered air.
  Arms: Filtered Air (FA)

SUMMARY:
The purpose of this research study to understand how environmental and genetic factors may be involved in lung function. Healthy Study participants will undergo a 1-day screening that includes a blood draw and breathing testing, return for a two-day series of testing to include blood draw, and brief breathing test before and after an inhaled challenge with either filtered air (FA) or ozone (O3). Participants return the next day for a brief breathing test, a blood draw and a procedure called bronchoscopy performed under conscious sedation to evaluate the lung after the challenge.

Participants then return 18 - 20 days later to repeat the two-day series of testing to be challenged with the exposure not received on the first series, (FA or O3). Each visit will take about 3 - 3.5 hours. Follow-up phone calls from the study team will occur at 24 hours after each 2-day test series. Total study duration is about one to one-and a half months.

DETAILED DESCRIPTION:
In brief, at V1 subjects will be assessed for baseline spirometry and venous blood analysis prior to exposure. The venous blood will be used to obtain PMNs for apoptosis assays, and serum for CFH and sCD163 levels. Additionally, this will be used to measure cytokines and growth factors. At each visit, if the subject is female, there will be a urine pregnancy test performed. Following this initial assessment, subjects will be challenged with FA or O3 and then spirometry will be performed, and venous blood will be obtained immediately following the exposure (V2). The subjects will then return 20 hours ±4h later for follow up studies (V3). There will be spirometry, a venous blood draw and urine pregnancy testing (if female) followed by bronchoscopy. At bronchoscopy, vital signs will be determined, including O2 sat. Patient then undergo an 18-20 day washout period before they are brought back in for V4 for the alternate challenge. This will follow the same protocol as outline above in the initial exposure and use the same series of analysis as the first set of visits. Therefore, we will fully characterize the biological response to ozone and filtered air in these same subjects.

ELIGIBILITY:
Inclusion Criteria

• Individuals between 18-35 yrs. of age (No subject will be excluded from the study on the basis of gender or ethnicity)

Exclusion Criteria

* Current smokers of tobacco products including e-cigarettes or those with previous smoking history within the prior 5 years
* Pregnant women and women who are presently lactating.
* Subjects that have received antibiotic administration or an upper respiratory infection within the previous 4 weeks
* College and graduate students or employees who are under direct supervision by any of the investigators in this protocol
* Alcohol or illicit substance abuse
* Chronic cardio/pulmonary respiratory disorders or other medical conditions as determined by the investigator
* Increased airway hyperresponsiveness at baseline as measured by a positive methacholine challenge response (methacholine PC20 FEV1 < 8 mg/ml)
* Subjects will be requested to refrain from antihistamines, nonsteroidal anti-inflammatory agents, antioxidants (e.g. beta-carotene, selenium, and lutein) and supplemental vitamins (e.g. C and E), for 1 week prior to, and during testing.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
change in ozone induced efferocytosis of lung macrophages (ability to clear dead or dying cells) | Baseline, 21 days
  Efferocytosis is defined by determining the number of apoptotic PMNs phagocytized by alveolar macrophages (BAL cytospins) versus the total number of macrophages ('efferocytic index')
Change in ozone induced phagocytosis of lung macrophages (ability to clear debris or bacteria) | Baseline, 21 days
  Bronchoalveolar macrophages are incubated with pHrodo™ dye-labeled particles. Macrophage phagocytosis will be defined by determining the number of macrophages that contain fluorescent particles versus the total macrophages Cell free hemoglobin and soluble CD163 - both are measured by commercial ELISA kit

SECONDARY OUTCOMES:
Change in ozone induced increase in cell free hemoglobin in bronchoalveolar lavage fluid and serum | Baseline, 21 days
  Measured by enzyme-linked immunosorbent assay (ELISA)
Change in ozone induced increase in soluble CD163 in bronchoalveolar lavage fluid and serum | Baseline, 21 days
  Measured by enzyme-linked immunosorbent assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tighe, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No